CLINICAL TRIAL: NCT00586716
Title: IVIG Treatment for Live-donor Renal Transplant Patients With a Positive Crossmatch and in Patients With High PRA
Brief Title: Intravenous Immune Globulin (IVIG) Treatment Protocol in Kidney Transplant Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54298
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 intravenous immune globulin (Other): Intravenous immunoglobulin for: patients who do not have a living donor, have a PRA greater than 30% for 3 consecutive months, and have one positive crossmatch with a cadaveric donor while on kidney transplant waiting list
  Interventions: Drug: intravenous immune globulin
- Group 2 intravenous immune globulin (Other): Intravenous immune globulin for patients who have living donors with positive crossmatch results.
  Interventions: Drug: intravenous immune globulin

INTERVENTIONS:
Drug: intravenous immune globulin — 0.5-2 gm/kg monthly (maximum dose of 140 gm/dose) x 4 treatments

SUMMARY:
The purpose of this study is to test the clinical and laboratory observations of IVIG therapy in the highly sensitized patient. We will study the effects of patients treated with IVIG or Cytogam in combination with plasmaphoresis to modulate the immune response in highly sensitized patients. The goal is to convert a positive crossmatch to a compatible crossmatch that would allow living related transplant to take place or to shorten time on the transplant waiting list.

DETAILED DESCRIPTION:
The purpose of this study is to test the clinical and laboratory observations of IVIG therapy in the highly sensitized patient. We will study the effects of patients treated with IVIG or Cytogam in combination with plasmaphoresis to modulate the immune response in highly sensitized patients. There are two arms in the study, one in which IVIG is administered to patients who have living donors with positive crossmatch results, and another in which intravenous immune globulin is administered to patients with no living donor and have a PRA greater than 30% for 3 consecutive months and a crossmatch with a cadaveric donor while on kidney transplant waiting list. The goal is to convert a positive crossmatch to a compatible crossmatch that would allow living related transplant to take place or to shorten time on the transplant waiting list.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* diagnosed with end stage renal disease
* currently receiving either hemodialysis or peritoneal dialysis
* active on the kidney or kidney/pancreas transplant list
* medical clearance of the kidney donor if live related transplant
* elevated panel reactive antibody (PRA) greater that 30% for 3 consecutive monthly tests and one positive crossmatch with a cadaveric donor while on the transplant waiting list

Exclusion Criteria:

* received IVIG within 6 months prior to enrollment
* HIV positive
* Positive Hepatitis Be-antigen and/or hepatitis B viral DNA
* Selective IgA deficiency or known antibodies to IgA
* Allergy to human immune globulin
* Pregnant or breast feeding

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-11; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Okechukwu Ojogho, MD, Principal Investigator — Loma Linda Universtiy Adventist Health Sciences Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Intravenous Immune Globulin no Living Donor: Patients who do not have a living donor, have a PRA greater than 30% for 3 consecutive months, and have one positive crossmatch with a cadaveric donor while on kidney transplant waiting list
  intravenous immune globulins : 0.5-2 gm/kg monthly (maximum dose of 140 gm/dose) x 4 treatments
- Group 2 Intravenous Immune Globulin With Living Donor: Patients who have living donors with positive crossmatch results.
  intravenous immune globulins : 0.5-2 gm/kg monthly (maximum dose of 140 gm/dose) x 4 treatments
Period: Overall Study
Arm/Group | Group 1 Intravenous Immune Globulin no Living Donor | Group 2 Intravenous Immune Globulin With Living Donor
Started | 14 | 8
Completed | 14 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IVIG no Living Donor: Intravenous immunoglobulin for: patients who do not have a living donor, have a PRA greater than 30% for 3 consecutive months, and have one positive crossmatch with a cadaveric donor while on kidney transplant waiting list
- IVIG With Living Donor: Intravenous immune globulin for patients who have living donors with positive crossmatch results.
- Total: Total of all reporting groups
Arm/Group | IVIG no Living Donor | IVIG With Living Donor | Total
Number analyzed (Participants) | 14 | 8 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 8 | 22
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Unknown | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Elimination of Donor Specific Antibodies
Time Frame: 1 year
Population: Study was terminated and no data for the outcome was collected/analyzed because it could not be located.
Groups:
- Intravenous Immune Globulin: Intravenous immune globulin for patients who have living donors with positive crossmatch results
Arm/Group | Intravenous Immune Globulin
Number analyzed (Participants) | 0

2. Secondary Outcome: Negative B and T Cell Crossmatch
Time Frame: 1year
Population: Study was terminated and no data for the outcome was collected/analyzed because it could not be located.
Arm/Group | Group 1 Intravenous Immune Globulin | Group 2 Intravenous Immune Globulin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Serious and non-serious adverse events were not collected/assessed.
Groups:
- Group 1 Intravenous Immune Globulin: Group 1 with Intravenous immune globulin with no living donor
- Group 2 Intravenous Immune Globulin: Group 2 intravenous immune globulin WITH living donor
Arm/Group | Group 1 Intravenous Immune Globulin | Group 2 Intravenous Immune Globulin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
A limitation to this study is early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes